CLINICAL TRIAL: NCT05988567
Title: Efficacy Testing of Melon Oil Olive Pressed Candy Products
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TCI Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 23-049-B
Record Dates: First submitted 2023-08-04; First posted 2023-08-14 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Skin Condition
MeSH Terms: conditions — Skin Diseases | interventions — Olive Oil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo candy (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo candy
- melon and oil olive pressed candy (Experimental)
  Interventions: Dietary Supplement: melon and oil olive pressed candy

INTERVENTIONS:
Dietary Supplement: Placebo candy — consume 2 tablets per day
  Arms: Placebo candy
Dietary Supplement: melon and oil olive pressed candy — consume 2 tablets per day
  Other Names: Melon, oil olive and pomegranate blend pressed candy
  Arms: melon and oil olive pressed candy

SUMMARY:
To assess melon and oil olive pressed candy on skin condition improvement

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged above 18 years old
* ITA° value 20°-41°

Exclusion Criteria:

* Involuntary subjects.
* Subjects who have a history of skin diseases such as psoriasis, eczema, atopic dermatitis, severe acne; or suffer from other chronic systemic disease.
* Those with known cosmetic, drug or food allergies.
* Female who is pregnant or nursing or planning to become pregnant during the course of the study.
* Subjects who have taken oral or topical corticosteroids and other anti-inflammatory drugs in the past 1 month.
* Use of any products or drugs that affect skin color such as fruit acid, salicylic acid (such as Hydroquinone preparations) in the past 2 months.
* In the past 3 months, the test site has used retinoic acid preparations or undergone chemical peeling, laser, pulse light and other medical aesthetic therapists
* Subjects who can not avoid long-term sun exposure

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-05-09 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
The change of skin wrinkles | Change from Baseline skin wrinkles at 12 weeks
  VISIA Complexion Analysis System was utilized to measure skin wrinkles. Units: arbitrary units
The change of skin texture | Change from Baseline skin texture at 12 weeks
  VISIA Complexion Analysis System was utilized to measure skin texture. Units: arbitrary units
The change of skin melanin index | Change from Baseline skin melanin index at 12 weeks
  Mexameter® MX18 was utilized to measure skin melanin index. Units: arbitrary units
The change of skin erythema index | Change from Baseline skin erythema index at 12 weeks
  Mexameter® MX18 was utilized to measure skin erythema index. Units: arbitrary units
The change of skin L* value | Change from Baseline L* value at 12 weeks
  Chroma Meter MM500 was utilized to measure skin L* value. Units: arbitrary units
The change of skin b* value | Change from Baseline b* value at 12 weeks
  Chroma Meter MM500 was utilized to measure skin b* value. Units: arbitrary units
The change of skin ITA° value | Change from Baseline ITA° value at 12 weeks
  Chroma Meter MM500 was utilized to measure skin ITA° value. Units: arbitrary units
The change of skin spots | Change from Baseline skin spots at 12 weeks
  VISIA Complexion Analysis System was utilized to measure skin spots. Units: arbitrary units
The change of skin UV spots | Change from Baseline skin UV spots at 12 weeks
  VISIA Complexion Analysis System was utilized to measure skin UV spots. Units: arbitrary units
The change of skin brown spots | Change from Baseline skin brown spots at 12 weeks
  VISIA Complexion Analysis System was utilized to measure skin brown spots. Units: arbitrary units

SECONDARY OUTCOMES:
The change of TEAC of blood | Change from Baseline TEAC at 12 weeks
  Venous blood was sampled to measure TEAC
The change of SOD of blood | Change from Baseline SOD at 12 weeks
  Venous blood was sampled to measure SOD
The change of GSH-Px of blood | Change from Baseline GSH-Px at 12 weeks
  Venous blood was sampled to measure GSH-Px

OTHER OUTCOMES:
The change of self-assessment skin and hair condition | Change from Baseline skin and hair condition at 12 weeks
  A self-assessment questionnaire was collected to evaluate skin and hair condition

CONTACTS AND LOCATIONS:
Overall Officials: Chia-Hua Liang, Prof., Principal Investigator — Chia Nan University of Pharmacy ＆ Science
Locations (1):
- Chia Nan University of Pharmacy & Science, Tainan, Taiwan

REFERENCES:
- [Derived] He Y, Bu Y, Chiang CF, Lin YH, Liang CH, Chan LP, Sun J. Multi-Plant Concentrated Powder Improved Skin Whitening: A Double-Blinded, Randomized, and Placebo-Controlled Clinical Study. J Cosmet Dermatol. 2025 Feb;24(2):e70011. doi: 10.1111/jocd.70011. PMID 39927597